CLINICAL TRIAL: NCT03140371
Title: An Evaluation of the Tolerance, Compliance and Acceptability of a Ready to Use, Liquid, High Energy, High Protein, Peptide-based Feed for Adults in Need of Nutrition Support - a Pilot Study
Brief Title: High Energy High Protein Peptide Feed Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HEHP16
Record Dates: First submitted 2017-02-21; First posted 2017-05-04 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Malnutrition; Malabsorption
Keywords: Enteral feeding; Oral nutritional supplements; Peptide-based feed; Hydrolysed feed; Semi-elemental feed
MeSH Terms: conditions — Malnutrition; Malabsorption Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High energy high protein peptide feed (Experimental): This is a one-arm study. Each patient recruited onto the study will receive the high energy, high protein peptide-based feed for a period of up to 4 weeks (28 days). The feed will be available as an enteral tube feed in a 500ml bottle, and as a Vanilla flavoured oral nutritional supplement in a 200ml plastic bottle. The appropriate feed presentation (tube feed or oral nutritional supplement) and prescription will be determined on an individual basis by the Dietitian responsible for the patient's nutritional management, based on the patient's clinical requirement and preference, and the Dietitian's clinical judgement.
  The study feed is classed as a 'Dietary Food for Special Medical Purposes' (EC Directive 1999/21/EC, 1999) .
  Interventions: Dietary Supplement: High energy high protein peptide feed study

INTERVENTIONS:
Dietary Supplement: High energy high protein peptide feed study — Each patient will receive the high energy, high protein peptide-based feed for a period of up to 4 weeks (28 days). The feed will be available as an enteral tube feed in a 500ml bottle, and as a Vanilla flavoured oral nutritional supplement in a 200ml plastic bottle. The appropriate feed presentation (tube feed or oral nutritional supplement) and prescription will be determined on an individual basis by the Dietitian responsible for the patient's nutritional management, based on the patient's clinical requirement and preference, and the Dietitian's clinical judgement.
  The study feed is classed as a 'Dietary Food for Special Medical Purposes' (EC Directive 1999/21/EC, 1999) .

SUMMARY:
Oral nutritional supplements and enteral tube feeds are commonly used to meet the nutritional requirements of patients with disease-related malnutrition, or who require medical nutrition support for other reasons. Some patients may not tolerate standard formulations containing whole proteins (typically due to maldigestion/malabsorption) leading to gastrointestinal symptoms (i.e. vomiting and diarrhoea). Without appropriate management, this may lead to reduced nutritional intake, increased nutritional losses and risk of malnutrition in patients who may already have elevated nutritional requirements due to their clinical conditions.

Poor tolerance to standard feed formulations can be managed with extensively hydrolysed (peptide-based) enteral feeds, where the protein source is provided in smaller proteins. Patients with elevated nutritional requirements, poor tolerance, maldigestion and/or malabsorption often require a higher energy, higher protein feed to meet their nutritional requirements in a smaller volume of feed.

The study feed is a high energy (1.5kcal/ml), high protein (7.5g protein/100ml) peptide-based feed, available as a 500ml enteral tube feed, and a 200ml Vanilla-flavour oral nutritional supplement. The study will investigate the gastrointestinal tolerance, compliance and acceptability of the high energy, high protein peptide-based feed in 60 adult patients requiring a peptide-based feed, in several NHS sites across England. Patients will be asked to take the study feed for 28 days. Data will be recorded using questionnaires with no invasive measures.

The primary outcome is gastrointestinal tolerance with secondary outcomes of compliance, acceptability, nutrient intake and anthropometry.

DETAILED DESCRIPTION:
Malnutrition or "undernutrition" in adults (≥18 years of age) is the deficiency of nutrients (energy, protein and micronutrients) which causes adverse effects on bodily composition, clinical and functional outcomes. Malnutrition can occur as a result of a number of factors including inadequate calorie intake, impaired nutrient absorption (malabsorption/maldigestion) or increased energy requirements usually associated with disease/illness e.g. cancer, inflammatory bowel disease and pancreatitis, and its management, e.g. chemotherapy and surgery. Patients who have or are at risk of malnutrition can be managed with a range of nutrition support strategies, including the use of oral nutritional supplements and enteral feeds (administered by feeding tubes such as nasogastric tubes, gastrostomies or jejunostomies). These feeds may provide either a sole source of nutrition or in combination with the diet.

A small group of patients requiring nutritional support experience severe malabsorption and maldigestion of nutrients (particularly protein and fat), resulting in them having an inadequate energy and nutrient supply. This may be due to inadequate functioning of the gastro-intestinal tract due to inflammation, reduced concentration of digestive enzymes and/or reduced surface area for nutrient absorption associated with some diseases and treatments. These may include patients with pancreatic enzyme deficiency (pancreatitis, pancreatic cancer, cystic fibrosis), inflammatory bowel disease, radiation enteritis and chemotherapy, short bowel syndrome, HIV-related gastrointestinal disorders, enteric fistulae or intolerance/allergy of unknown cause. Some of these patients will not be able to tolerate a standard feed containing whole protein and fat. In these cases oral nutritional supplements and enteral tube feeds known as 'extensively hydrolysed', 'semi-elemental' or 'peptide-based' with extensively digested protein (containing peptides and small proteins) and containing more easily absorbed types of fat (medium chain triglycerides (MCTs)), can help improve digestion and absorption.

Peptide-based feeds have been used effectively in the dietary management of patients with Crohn's disease, pancreatitis, pancreatectomy, radiation enteritis and chemotherapy, HIV-related GI disorders and short bowel syndrome. The use of MCTs in patients with fat (long chain triglyceride (LCT)) malabsorption has been shown to decrease steatorrhoea, decrease dyspepsia and improve nutritional status. Feed formulations with a mixture of MCTs and LCTs are also thought to provide beneficial effects.

Such specialised, ready to use feeds have been commonly used in clinical practice for many years. However, the energy density (1kcal/ml) and the protein content (4g/100ml) of some such feeds have meant that patients are often unable to tolerate the required volumes of feed either orally or via tube to meet their nutritional requirements, which are often elevated by their disease. Therefore, in order to meet the nutritional requirements of patients with poor feed tolerance, a more energy dense (1.5kcal/ml), higher protein (7.5g protein/100ml), nutritionally complete peptide-based feed for oral and tube feeding may be required.

The study feed is a high energy (1.5kcal/ml), high protein (7.5g protein/100ml) peptide-based feed, available as a 500ml enteral tube feed, and a 200ml Vanilla-flavour oral nutritional supplement. However, the tolerance, compliance and acceptability of this feed is unknown in this patient group who have complex clinical conditions. Therefore this study is required to assess gastrointestinal tolerance, compliance and acceptability of this high energy density (1.5kcal/ml), high protein (7.5g/100ml), peptide-based feed in community patients requiring nutrition support in clinical practice.

60 adult patients requiring a peptide-based feed will be recruited from several NHS sites across England. Patients will be asked to take the study feed for 4 weeks (28 days), in a quantity advised by their Dietitian. Data will be recorded at baseline, Week 4 and throughout the study using questionnaires with no invasive measures.

The primary outcome is gastrointestinal tolerance with secondary outcomes of compliance to prescribed study feed volumes, acceptability of the study feed, nutrient intake and anthropometry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 years and over
* Requiring a peptide-based feed to meet nutritional requirements
* Expected to receive at least 300kcal if taken orally or at least 500kcal if taken by tube

Exclusion Criteria:

* Patients receiving total parenteral nutrition
* Patients with major hepatic dysfunction (i.e. decompensated liver disease)
* Patients with major renal dysfunction (i.e. requiring filtration or Stage 4/5 chronic kidney disease (CKD))
* Patients in intensive care
* Patients with galactosaemia or severe lactose intolerance
* Participation in other clinical studies within 2 weeks prior to entry of this study
* Investigator concern around willingness/ability of patient to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Gastro-intestinal tolerance (change is assessed at different timepoints) | To be completed on Days 1, 2, 3, 7, 14, 21, 26, 17 and 28
  Questionaire detailing any GI symptoms, severity and change from usual

SECONDARY OUTCOMES:
Compliance with feed prescription | 28 days
  Brief questionnaire on amounts offered and amounts actually consumed, compared to recommended amount.
Acceptability | 1 day (Day 28)
  Brief tick-box questionnaire on overall liking and acceptability of product
Weight (change will be assessed at different timepoints) | To be completed at Baseline and Day 28 (2 days)
  Measurements of weight (kg) at baseline and end of study
Height (change will be assessed at different timepoints) | To be completed at Baseline and Day 28 (2 days)
  Measurements of height (cm) at baseline and end of study
Nutrient intake | To be completed at Baseline and Day 28 (2 days)
  24hr dietary recall at baseline and end of study, subsequently analysed in dietary software.
Patient history | To be completed at Baseline (Day 1)
  A detailed patient history will be recorded at baseline

CONTACTS AND LOCATIONS:
Locations (10):
- United Kingdom (10):
  - Cumbria Partnership NHS Foundation Trust, Whitehaven, Cumbria
  - Derby Teaching Hospitals NHS Foundation Trust, Derby, Derbyshire
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester, Gloucestershire
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford, Lonodn
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Frimley Health NHS Foundation Trust, Frimley
  - Guys and St Thomas NHS Foundation Trust, London
  - Lewisham and Greenwich NHS Foundation Trust, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Great Western Hospitals NHS Foundation Trust, Swindon

IPD SHARING:
Plan to Share IPD: No